CLINICAL TRIAL: NCT02324348
Title: Impact of Immediate Stent Implantation Versus Deferred Stent Implantation on Infarct Size and Microvascular Perfusion in Patients With ST-segment Elevation Myocardial Infarction
Brief Title: Efficacy and Safety Study of Deferred Stenting in Patients With STEMI
Acronym: INNOVATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Cheol Woong Yu, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-3
Record Dates: First submitted 2014-08-26; First posted 2014-12-24 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate coronary stenting (Placebo Comparator): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, stent implantation is done on the initial procedure in immediate coronary stenting group
  Interventions: Procedure: Immediate coronary stenting
- Deferred coronary stenting (Active Comparator): Within enrolled patients who agreed to participate in the study, signed informed consent and being satisfied with inclusion and exclusion criteria, only TIMI Ⅲ flow achievement is done on the initial procedure and stent implantation is deferred after 5-7 days admission in the deferred coronary stenting group.
  Interventions: Procedure: Deferred coronary stenting

INTERVENTIONS:
Procedure: Deferred coronary stenting — Abciximab (0.25㎎/㎏) intracoronary injection will be performed to all possible patients after guidewire has passed culprit lesion. Additional manual thrombus aspiration or balloon angioplasty can be performed by operator to achieve TIMI Ⅲ flow. When TIMI Ⅲ flow is achieved after these procedures, patient will be randomized to immediate stenting or deferred stenting group. In deferred stenting group, second stage procedure (stent implantation) will be done at 5 to 7 days after TIMI Ⅲ flow has achieved.
  Arms: Deferred coronary stenting
Procedure: Immediate coronary stenting — Abciximab (0.25㎎/㎏) intracoronary injection will be performed to all possible patients after guidewire has passed culprit lesion. Additional manual thrombus aspiration or balloon angioplasty can be performed by operator to achieve TIMI Ⅲ flow. When TIMI Ⅲ flow is achieved after these procedures, patient will be randomized to immediate stenting or deferred stenting group. In immediate stenting group, stenting will be done immediate after achieving TIMI III flow during initial procedure.
  Arms: Immediate coronary stenting

SUMMARY:
It is known that no reflow phenomenon by microvascular obstruction after revascularization in STEMI increase infarct size, cardiac remodeling, and a risk of late mortality. Major mechanism of microvascular obstruction is distal embolization during procedure. Some investigators showed deferred stenting decreased the degree of microvascular obstruction compared with immediate stenting in STEMI. The aim of current study is to compare impact of immediate stent implantation versus deferred stent implantation on infarct size and microvascular perfusion in patients with ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
1. Patients will be enrolled if they agree to participate in the study and sign informed consent among patients who are satisfied with inclusion and exclusion criteria. Acceptance of the study will be taken concurrently at the situation when the patient admitted via emergency department with the diagnosis of STEMI and informed consent of primary coronary angiography and intervention is taken. Considering emergent situation of the procedure, it is thought to be impossible to take informed consent of the study before procedure and after achieving TIMI flow. Duty operator will inform to the patient when taking informed consent of primary coronary angiography and intervention that the patient will be randomized to immediate coronary stenting group or deferred coronary stent group, and explain about theoretical background of deferred coronary stenting. To all patients, aspirin 300㎎, clopidogrel 600㎎ are administered orally and heparin intravenously until achieving ACT (activated clotting time) between 200 and 250 seconds. Maximal total dose of unfractionated heparin of 100 unit/㎏ will be administered before intervention.
2. Transradial or transfemoral approach will be determined on operator's decision. Flow of the infarct related artery (IRA) will be checked as total occlusion, TIMI 0, Ⅰ or Ⅱ after coronary angiography.
3. Abciximab (0.25㎎/㎏) intracoronary injection will be performed to all possible patients after guidewire has passed culprit lesion. Additional manual thrombus aspiration or balloon angioplasty can be performed by operator to achieve TIMI Ⅲ flow. When TIMI Ⅲ flow is achieved after these procedures, patient will be randomized to immediate stenting or deferred stenting group.
4. Although stent implantation without balloon angioplasty is preferred in immediate stenting group, balloon angioplasty can be performed to achieve distal flow. In deferred stenting group, second stage procedure (stent implantation) will be done at 5 to 7 days after TIMI Ⅲ flow has achieved.
5. On coronary intervention (stent implantation), all possible cases will be implanted with Nobori Biolimus A9-eluting coronary stent (Terumo, Tokyo, Japan). (Other stents can be used if the length of the lesion cannot be covered with Nobori stent.)
6. In both group, abciximab continuous intravenous infusion on a dose of 0.125 ㎍/㎏/min (maximum dose 10 ㎍/min) will be done after initial procedure if possible. (Intracoronary injection and intravenous infusion of abciximab should be done unless there is no contraindication of abciximab.)
7. In both group, subcutaneous enoxaparin (low molecular weight heparin) injection will be done twice daily until 3 days after procedure if possible. In case of stent implantation in the fifth to seventh day within deferred coronary stenting group, enoxaparin injection can be extended until deferred intervention.
8. Transradial and transfemoral approach are all possible. If procedure is done with transfemoral approach, sheath removal will be done after continuous intravenous abciximal infusion of 12 hours and enoxaparin injection after hemostasis has been confirmed.
9. In case of residual stenosis of IRA is below 30% within deferred coronary stenting group, intravascular ultrasonography (IVUS) will be performed at the secondary procedure and withdrawal of stenting can be done upon operator's discretion.
10. In case of multivessel disease, intervention of non-IRA will be deferred in both groups. Therefore, PCI on IRA and non-IRA will be done concurrently in deferred coronary stenting group.
11. Patient will maintain dual antiplatelet therapy of aspirin 100㎎ and clopidogrel 75㎎ after PCI.
12. Among prescribed drugs after PCI, statin agent can be used upon operator's discretion.
13. Cardiac MRI is done on the period of 30±7 days after diagnosed as STEMI in both group.
14. Follow-up period is 1 month ± 1 week, 6 month ± 4 week, and 12 month ± 4 week in both group. Transthoracic echocardiography will be done at 6 month ± 4 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* more than 30 minutes of duration of typical chest pain
* 1mm or more of ST elevation on 2 or more continuous leads
* chest pain within 12 hours
* Thrombolysis In Myocardial Infarction (TIMI) flow 0, Ⅰ or Ⅱ before procedure
* TIMI Ⅲ flow after balloon angioplasty, intracoronary abciximab infusion, or thrombus aspiration
* accepted informed consent

Exclusion Criteria:

* cardiogenic shock
* previous history of myocardiac infarction, or coronary artery bypass graft
* rescue percutaneous coronary intervention after fibrinolysis
* life expectancy < 1 year
* left main disease (included if left main lesion is not infarct related artery)
* contraindication to cardiac MRI
* STEMI due to stent thrombosis
* anticipated risk of acute closure when assigned as deferred stenting group in the condition major dissection (type C~F) has occurred during procedure achieving TIMI flow involving balloon angioplasty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Infarct size measured by cardiac magnetic resonance image (MRI) | Post MI 30 days

SECONDARY OUTCOMES:
Microvascular obstruction (MVO) volume measured by cardiac MRI | Post MI 30 days
Ratio of MVO volume to infarct size | Post MI 30 days
Enzymatic infarct size | Post MI 30 days
Degree of resolution of ST-segment elevation | 1 hour after coronary stenting
CTFC (corrected TIMI frame count) | Immediately after coronary stenting
Myocardial brush grade | Immediately after coronary stenting
Rate of slow flow or no reflow phenomenon (TIMI flow≤2) | Immediately after coronary stenting

OTHER OUTCOMES:
Left ventricle (LV) ejection fraction | Post MI 6 months
Left ventricle (LV) remodelling index | Post MI 6 months
MACCE (major adverse cardiac and cerebrovascular event) | Post MI 1, 6, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Woong Yu, M.D.,Ph.D., Principal Investigator — Cardiovascular center, Korea university Anam hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kook H, Lee HJ, Kim MN, Yu CW, Kim JS, Joo HJ, Park JH, Hong SJ, Kim TH, Jang HJ, Park JS, Choi RK, Choi YJ, Kim YM, Lim DS, Ro YM. Effects of deferred versus immediate stenting on left ventricular function in patients with ST elevation myocardial infarction. Medicine (Baltimore). 2021 Jul 16;100(28):e26598. doi: 10.1097/MD.0000000000026598. PMID 34260542
- [Derived] Kim JS, Lee HJ, Woong Yu C, Kim YM, Hong SJ, Park JH, Choi RK, Choi YJ, Park JS, Kim TH, Jang HJ, Joo HJ, Cho SA, Ro YM, Lim DS. INNOVATION Study (Impact of Immediate Stent Implantation Versus Deferred Stent Implantation on Infarct Size and Microvascular Perfusion in Patients With ST-Segment-Elevation Myocardial Infarction). Circ Cardiovasc Interv. 2016 Dec;9(12):e004101. doi: 10.1161/CIRCINTERVENTIONS.116.004101. PMID 27965296